CLINICAL TRIAL: NCT03869684
Title: A Double-Masked, Randomized, Multicenter, Placebo-Controlled, Parallel-Group Study to Assess the Safety, Tolerability, and Efficacy of MT-0814 for the Treatment of Patients With Age-Related Macular Degeneration
Brief Title: A Study to Assess the Safety, Tolerability and Effectiveness of MT-0814 for the Treatment of Age-related Macular Degeneration
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study terminated for safety reasons
Sponsor: Senju Pharmaceutical Co., Ltd. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-0814/2-01
Record Dates: First submitted 2019-03-01; First posted 2019-03-11 (Actual); Results first posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-03

CONDITIONS: Age-related Macular Degeneration
Keywords: Exudative; Wet; AMD; Age-related macular degeneration; Age related macular degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MT-0814 High dose (Experimental)
  Interventions: Drug: MT-0814
- MT-0814 Low dose (Experimental): MT-0814 plus placebo
  Interventions: Drug: MT-0814; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT-0814 — Randomly assigned dose
  Arms: MT-0814 High dose; MT-0814 Low dose
Drug: Placebo — Placebo manufactured to mimic MT-0814
  Arms: MT-0814 Low dose; Placebo

SUMMARY:
Age-related macular degeneration (AMD) is the leading cause of blindness among adults in North America. The current standard of care for patients with exudative ("wet") AMD is anti-vascular endothelial growth factor (anti-VEGF) therapy which must be administered by an injection into the eye every 4-8 weeks. MT-0814 is being developed for the treatment of patients with exudative AMD, and could offer an alternative, safer and less burdensome therapy.

ELIGIBILITY:
Inclusion Criteria:

* Must agree to sign informed consent form, and to comply with protocol requirements, including study visits.
* Must have clear optic media in the study eye that is capable of producing high-quality fundus images.

Exclusion Criteria:

* Has active CNV due to causes other than AMD in the study eye.
* Has retinal vascular disease or retinal degeneration other than AMD in the study eye.
* Has had intraocular surgery, cataract surgery or LASIK surgery on the study eye within 90 days prior to the study.
* Has had yttrium aluminum garnet (YAG) laser capsulotomy on the study eye within 30 days prior to the study.
* Has active inflammation, infection, or other severe ocular disease in either eye.
* Has aphakia in the study eye.
* Has uncontrolled glaucoma or a history of previous glaucoma filter surgery in either eye.
* Is a contact lens wearer and is unable to discontinue their use in both eyes for the duration of the study.
* Has a serious allergy to, or experienced a prior significant adverse reaction to fluorescein angiography (FA) or indocyanine green angiography (ICGA).
* Has participated in any other clinical trial and/or has taken any investigational drug or product within 90 days prior to the study.

Other protocol-defined inclusion/exclusion criteria could apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-04-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Senju Investigational Site, Peoria, Arizona
  - Senju Investigational Site, Phoenix, Arizona
  - Senju Investigational Site, Pasadena, California
  - Senju Investigational Site, Redlands, California
  - Senju Investigational Site, Altamonte Springs, Florida
  - Senju Investigational Site, Clearwater, Florida
  - Senju Investigational Site, Melbourne, Florida
  - Senju Investigational Site, Tallahassee, Florida
  - Senju Investigational Site, Arlington, Texas
  - Senju Investigational Site, Houston, Texas
  - Senju Investigational Site, San Antonio, Texas
  - Senju Investigational Site, The Woodlands, Texas
  - Senju Investigational Site, Murray, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | MT-0814 Low Dose | MT-0814 High Dose
Started | 3 | 5 | 5
Completed | 1 | 2 | 2
Not Completed | 2 | 3 | 3
Not completed — Adverse Event | 0 | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Study prematurely terminated by sponsor | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MT-0814 Low Dose | MT-0814 High Dose | Total
Number analyzed (Participants) | 3 | 5 | 5 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 0 | 3
  >=65 years | 1 | 4 | 5 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 2 | 8
  Male | 1 | 1 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 5 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Whte | 3 | 5 | 5 | 13
  Other | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 5 | 13
Best-corrected Visual Acuity (BCVA) : Study eye [Mean (Standard Deviation); unit: Letters] — BCVA was measured using an eye chart and is reported as number of letters read correctly using Early Treatment of Diabetic Retinopathy Study (ETDRS) Scale (0 to 100 letters) in study eye. Lower number of letters read correctly, worse the vision.
  Study eye: eye that meets inclusion criteria. If both eyes meet all inclusion and exclusion criteria, the eye with the lower BCVA at Screening will be selected as the study eye. If both eyes meet all inclusion criteria and have identical BCVA at Screening, selection of the study eye will be at the investigator's discretion.
  Letters | 62.0 (10.82) | 66.8 (7.98) | 71.2 (4.15) | 67.4 (7.74)
Central Subfield Thickness (CSFT) : Study eye [Mean (Standard Deviation); unit: mm] | 0.2990 (0.04015) | 0.3748 (0.05981) | 0.3954 (0.08581) | 0.3652 (0.07369)

OUTCOME MEASURES:

1. Primary Outcome: Change in Best-corrected Visual Acuity (BCVA) : Study Eye
Description: Change from Baseline in BCVA. BCVA was measured using an eye chart and is reported as number of letters read correctly using Early Treatment of Diabetic Retinopathy Study (ETDRS) Scale (0 to 100 letters) in study eye. Lower number of letters read correctly, worse the vision.
  Study eye: eye that meets inclusion criteria. If both eyes meet all inclusion and exclusion criteria, the eye with the lower BCVA at Screening will be selected as the study eye. If both eyes meet all inclusion criteria and have identical BCVA at Screening, selection of the study eye will be at the investigator's discretion.
Time Frame: Baseline and Week 12
Population: Full-analysis set (FAS): The FAS consisted of all participants who were randomly assigned to receive double-masked study drug and who have received at least 1 dose of study drug. All analyses using the FAS grouped participants according to randomly assigned treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: letters
Arm/Group | Placebo | MT-0814 Low Dose | MT-0814 High Dose
Number analyzed (Participants) | 3 | 5 | 5
letters | 0.4 [-7.7 to 8.5] | 0.3 [-5.6 to 6.1] | 0.1 [-6.1 to 6.3]

2. Secondary Outcome: Change in Central Subfield Thickness (CSFT) : Study Eye
Description: Change from Baseline in CSFT, measured by Optical Coherence Tomography (OCT).
  Study eye: eye that meets inclusion criteria. If both eyes meet all inclusion and exclusion criteria, the eye with the lower BCVA at Screening will be selected as the study eye. If both eyes meet all inclusion criteria and have identical BCVA at Screening, selection of the study eye will be at the investigator's discretion.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Placebo | MT-0814 Low Dose | MT-0814 High Dose
Number analyzed (Participants) | 3 | 5 | 5
mm | -0.0053 [-0.0628 to 0.0523] | -0.0016 [-0.0412 to 0.0380] | 0.0026 [-0.0387 to 0.0438]

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Adverse events were analyzed in terms of Treatment-Emergent Adverse Events (TEAEs), which were defined as any event not present before exposure to study drug or any event already present that worsened in either intensity or frequency after exposure to the study drug.
Arm/Group | Placebo | MT-0814 Low Dose | MT-0814 High Dose
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5 | 2/5
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=3) | MT-0814 Low Dose (N=5) | MT-0814 High Dose (N=5)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=3) | MT-0814 Low Dose (N=5) | MT-0814 High Dose (N=5)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract nuclear (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neovascular age-related macular degneration (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Subretinal fluid (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Mitral valve prolapse (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (2)
Dry age-related macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tension headach (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
High density lipoprotein decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
All of the efficacy and safety measurements applied in this study are widely used and generally recognized as reliable, accurate, and relevant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-29): https://cdn.clinicaltrials.gov/large-docs/84/NCT03869684/Prot_SAP_000.pdf